CLINICAL TRIAL: NCT00337389
Title: A Phase III Multi-Center Randomized Clinical Trial to Evaluate the Safety and Efficacy of CoFactor and 5-Fluorouracil (5-FU) Plus Bevacizumab Versus Leucovorin and 5-FU Plus Bevacizumab as Initial Treatment for Metastatic Colorectal Carcinoma
Brief Title: Phase III Randomized Study of 5-FU, CoFactor, and Avastin vs. 5-FU, LV and Avastin for First-Line Colorectal Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mast Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 510-05
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Metastatic Colorectal Cancer; Colon Cancer; Rectal Cancer
Keywords: Metastatic; Colorectal; Cancer; CoFactor; Stage IV
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; 5,11-methenyltetrahydrohomofolate

ARMS (2):
- 1 (Experimental): CoFactor, 5-FU, Avastin
  Interventions: Drug: 5- Fluorouracil (5-FU); Drug: bevacizumab (Avastin); Drug: CoFactor (ANX-510)
- 2 (Active Comparator): Leucovorin, 5-FU, Avastin
  Interventions: Drug: 5- Fluorouracil (5-FU); Drug: bevacizumab (Avastin); Drug: Leucovorin

INTERVENTIONS:
Drug: 5- Fluorouracil (5-FU)
Drug: bevacizumab (Avastin)
Drug: Leucovorin
  Arms: 2
Drug: CoFactor (ANX-510)
  Arms: 1

SUMMARY:
To compare the progression-free survival time (PFS) in patients treated with 5-FU modulated with CoFactor (plus bevacizumab) to 5-FU modulated with leucovorin (plus bevacizumab) in patients with Metastatic Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Greater or equal to 18 years of age.
2. Surgically incurable, metastatic disease from proven colon or rectal adenocarcinoma.
3. Life expectancy of at least 3 months.
4. Histologically confirmed metastatic disease. Histological confirmation may be waived if needle biopsy presents a significant risk to the subject and the clinical setting is clinically consistent with metastasis of colorectal cancer, e.g. surgical findings at laparotomy, or positive PET scan, synchronous histologically confirmed primary tumor with typical metastatic pattern (stage D disease). Waiver can only be granted by the Sponsor, and these cases will be kept to less than 10% of the total study population.
5. Measurable disease. At least one unidimensionally measurable lesion with a diameter ≥10 mm using spiral CT scans (use of spiral CT must be documented in medical records and used consistently throughout the study) or ≥20 mm using conventional CT or MRI scans.
6. No prior systemic chemotherapy or immunotherapy for metastatic or advanced local disease. However patients may have had radiosensitizing doses of fluoropyrimidines (only 5-FU or capecitabine, with or without leucovorin or levamisole is permitted) if completed 6 months prior to treatment on this protocol. No prior irinotecan or oxaliplatin in combination with radiotherapy is allowed.
7. Prior adjuvant therapy is allowed if completed more than 6 months prior to treatment on this protocol. Regimens which included oxaliplatin and irinotecan are allowed.
8. ECOG Performance Status is 0-2 or Karnofsky performance level of 100-70.
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Any prior exposure to bevacizumab.
2. A known intolerance to fluoropyrimidine (5-FU, capecitabine, floxuridine, UFT) therapy suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency.
3. Use of the following drugs are not permitted on the protocol: sorivudine (or other nucleoside analogue), or Brivudin™ (or other DPD inhibitor).
4. Pregnancy or lactation. Women with a positive (or no) serum or urine pregnancy test within 15 days of Cycle 1 Week 1. Women must have been amenorrheic for at least 12 consecutive months to be considered to lack potential for child bearing.
5. If sexually active and of child-bearing potential, failure to agree to use adequate contraception during this study and for 60 days after discontinuation of study medication.
6. A concurrent infection, including diagnoses of FUO and evidence of possible central line sepsis (subjects must be afebrile at the start of therapy).
7. Any unstable oncologic emergency syndromes: superior vena cava syndrome, rising bilirubin needing stent placement, spinal cord compression, active bleeding, etc.
8. History of CNS metastasis, or other brain tumor, or history of stroke.
9. Radiation therapy within 6 weeks of Cycle 1 Week 1, or any radiation therapy which encompasses target lesions selected for this study unless those lesions have documented progression of disease.
10. Major surgery, open biopsy, or significant traumatic injury within 4 weeks of Cycle 1 Week 1, or anticipated need for major surgical procedure during the course of the study.
11. Fine needle aspiration or placement of a central line catheter within 7 days of Cycle 1 Week 1.
12. Inadequate bone marrow, liver or kidney function defined as:

    * Serum creatinine more than 1.5 times the upper limit of normal,
    * Urine protein to creatinine ratio >1,
    * Serum bilirubin > 2 times the upper limit of normal,
    * ANC < 1.5 x 109/L,
    * Hemoglobin < 9.0 g / dL
    * Platelet count < 90 x 109/L,
    * SGOT (AST) and SGPT (ALT) more than 3 times the upper limit of normal, or more than 5 times the upper limit of normal for subjects with documented liver metastases.
13. Myocardial infarction, transient ischemic attack, cerebral bleeding, translumenal cardiac angiography or cardiac stent placement or other arterial thrombotic event within 12 months prior to Cycle 1 Week 1.
14. Active, clinically significant cardiovascular or symptomatic arterial peripheral vascular disease [e.g., uncontrolled hypertension, congestive heart failure, claudication, unstable angina, symptomatic cardiac arrhythmia, or New York Heart Association (NYHA) Class 2 or greater].
15. Presence of serious non-healing wounds, gastro-duodenal ulcers active by endoscopy, gastro-intestinal perforation or intra-abdominal abscess, skin ulcers, or bone fractures.
16. INR >1.5 unless on therapeutic doses of oral anticoagulants (e.g. warfarin). If so, must have an in-range INR (usually between 2-3) on a stable dose of drug.
17. Participation in another experimental drug study within 4 weeks prior to Cycle 1 Week 1.
18. Known or suspected anaphylaxis reaction to leucovorin or any allergic reaction to a drug which, in the opinion of the Investigator, suggests an increased potential for a hypersensitivity to CoFactor or other study drug including excipients.
19. Presence of organ allograft requiring immunosuppressive therapy.
20. Unwilling or unable to comply with the study protocol or history of psychiatric disability judged by the investigator to preclude granting of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Progression Free Survival

SECONDARY OUTCOMES:
Response Rate
Overall Survival
Incidence and Severity of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: M. Wasif Saif, MD, MBBS, Study Chair — Yale University
Locations (47):
- United States (46):
  - Research Center In, Florence, Alabama
  - Research Center In, Anaheim, California
  - Research Center In, Apple Valley, California
  - Research Center In, Beverly Hills, California
  - Research Center In, Irvine, California
  - Research Center In, Mission Hills, California
  - Research Center In, Poway, California
  - Research Center In, Rancho Mirage, California
  - Mercy General Hospital, Sacramento, California
  - Research Center In, Sacramento, California
  - Research Center In, San Diego, California
  - Research Site In, San Diego, California
  - Research Center In, Vista, California
  - Research Center In, Boynton Beach, Florida
  - Research Center In, Merritt Island, Florida
  - Research Center In, Port Saint Lucie, Florida
  - Research Center In, Tarpon Springs, Florida
  - Research Center In, Gurnee, Illinois
  - Research Center In, Joliet, Illinois
  - Research Center In, Skokie, Illinois
  - Research Center In, Indianapolis, Indiana
  - Research Center In, Wichita, Kansas
  - Research Center In, Hazard, Kentucky
  - Research Center In, Baltimore, Maryland
  - Research Center In, Flint, Michigan
  - Research Center In, Free Soil, Michigan
  - Research Center In, Grand Rapids, Michigan
  - Research Center In, Port Huron, Michigan
  - Research Center In, Jackson, Mississippi
  - Research Center In, Henderson, Nevada
  - Research Center In, Las Vegas, Nevada
  - Research Center In, Reno, Nevada
  - Research Center In, Cherry Hill, New Jersey
  - Research Center In, Farmington, New Mexico
  - Research Center In, East Setauket, New York
  - Research Center In, Greenville, North Carolina
  - Research Center In, Middletown, Ohio
  - Research Center In, Cranston, Rhode Island
  - Research Center In, Charleston, South Carolina
  - Research Center In, Columbia, South Carolina
  - Research Center In, Chattanooga, Tennessee
  - Research Center In, Collierville, Tennessee
  - Research Center In, Fort Worth, Texas
  - Research Center In, Ogden, Utah
  - Research Center In, Lacey, Washington
  - Research Center In, Walla Walla, Washington
- Research Center In, Zrenjanin, Serbia and Montenegro